CLINICAL TRIAL: NCT03505385
Title: Effects of a Unique Co-created Intervention With Care Home Residents and University Students Following a Service-learning Methodology to Reduce Sedentary Behaviour.
Acronym: GET READY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glasgow Caledonian University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 747490
Record Dates: First submitted 2018-04-12; First posted 2018-04-23 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2019-08

CONDITIONS: Physical Activity; Sedentary Behaviour; Care Home Residents
Keywords: Co-creation; Service-learning methodology
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Co-created intervention (Experimental): The Get Ready (GR) intervention was delivered one-to-one with the care home resident and a relevant family member during a 12-week period:
  1. The familiarisation stage aimed to build a rapport with two long-term achievement goals to sit less and move more with the resident and the family member and consisted of two sessions, one in week 1 (50-60minutes) and the other in week 3 (30-40 minutes).
  2. The ramping up stage aimed to review the rapport and reach an achievable consensus with the resident and the family member. It consisted of two sessions, one in week 5 and the other in week 7 (20-30 minutes each).
  3. The maintenance stage aimed at integrating behaviours and included two sessions, one in week 9 and the other at week 12 (20-30 minutes each). Sessions 5 and 6 were used to understand how the resident was getting on with their short-term GR goals, facilitating some problem-solving discussions.
  Interventions: Behavioral: Co-created intervention - Get Ready (GR)
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Co-created intervention - Get Ready (GR) — The Get Ready (GR) intervention was delivered one-to-one with the care home resident and a relevant family member during a 12-week period:
  1. The familiarisation stage aimed to build a rapport with two long-term achievement goals to sit less and move more with the resident and the family member and consisted of two sessions, one in week 1 (50-60minutes) and the other in week 3 (30-40 minutes).
  2. The ramping up stage aimed to review the rapport and reach an achievable consensus with the resident and the family member. It consisted of two sessions, one in week 5 and the other in week 7 (20-30 minutes each).
  3. The maintenance stage aimed at integrating behaviours and included two sessions, one in week 9 and the other at week 12 (20-30 minutes each). Sessions 5 and 6 were used to understand how the resident was getting on with their short-term GR goals, facilitating some problem-solving discussions.
  Arms: Co-created intervention

SUMMARY:
Background. There is a growing demand for long-term care settings. Care-home residents are a vulnerable group with high levels of physical dependency and cognitive impairment. Long-term care facilities' policy need to adapt and offer more effective and sustainable interventions to address their complex physical and mental health needs. Despite the increasing emphasis on patient and public involvement, marginalised groups such as care-home residents, can be overlooked when including people in the research process. The GET READY project aims to integrate service-learning methodology into Physical Therapy and Sport Sciences University degrees by offering students individual service opportunities (placements) with residential care homes, in order to co-create the best suited intervention with researchers, older adults of both genders (end-users) in care homes, health professionals, caregivers, family members and policy makers.

Methods. Stage 1 will integrate a service-learning methodology within a Physical Therapy module in Glasgow and Sport Sciences module in Barcelona, design two workshops for care home residents and conduct a co-creation protocol. Stage 2 will assess the intervention feasibility, safety and preliminary effects of the co-created intervention in a group of 33 care home residents, within a two-armed pragmatic randomized clinical trial.

ELIGIBILITY:
Inclusion Criteria:

- Care Home residents ≥ 70 years old.

Exclusion Criteria:

* Comorbidity preventing participation (e.g. severe breathlessness, pain, or severe neurological disease).
* Life expectancy of less than one year.
* Being unlikely to undertake the intervention regularly.
* Severe dementia.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Change in minutes spent in sedentary behaviour | During 7 days. Outcome measure will be collected at baseline and at the end of the intervention (up to 24 weeks)
  Number of minutes spent in activities requiring ≤ Metabolic Equivalent Tasks with ActivPal monitor.
Change in sitting time | During 7 days. Outcome measure will be collected at baseline and at the end of the intervention (up to 24 weeks).
  Number of minutes spent in a sitting position with ActivPal monitor.

SECONDARY OUTCOMES:
Change in health-related quality of life | Outcome measure will be collected at baseline and at the end of the intervention (up to 24 weeks).
  EuroQoL - 5D
Physical Function | Outcome measure will be collected at baseline and at the end of the intervention (up to 24 weeks).
  Short Physical Performance Battery

CONTACTS AND LOCATIONS:
Locations (1):
- The Erskine Glasgow Home, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gine-Garriga M, Sandlund M, Dall PM, Chastin SFM, Perez S, Skelton DA. A co-created intervention with care home residents and university students following a service-learning methodology to reduce sedentary behaviour: The GET READY project protocol. J Frailty Sarcopenia Falls. 2018 Sep 1;3(3):132-137. doi: 10.22540/JFSF-03-132. eCollection 2018 Sep. PMID 32300702